CLINICAL TRIAL: NCT04406597
Title: Safety, Effectiveness and Operability of Using the New Tissue Containment System With Hard Pipes Which Can Assemble With Detachable Trocars Seamlessly for Tissue Removal During Laparoscopic Ovarian Cystectomy
Brief Title: Safety, Effectiveness and Operability of Using the New Tissue Containment System During Laparoscopic Ovarian Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jing Liang, Vice Director of Obstetrics and Gynecology, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTCS-LOC
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Ovary Neoplasm; Surgery
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the New Tissue Containment System group (Experimental): Using the New Tissue Containment System during Laparoscopic Ovarian Cystectomy
  Interventions: Device: the New Tissue Containment System
- Open group (No Intervention): Without any protection system during Laparoscopic Ovarian Cystectomy

INTERVENTIONS:
Device: the New Tissue Containment System — Laparoscopic Ovarian Cystectomy using the New Tissue Containment System
  Arms: the New Tissue Containment System group

SUMMARY:
The study is designed to evaluate the safety, effectiveness and operability of performing in-bag cystectomy and morcellation with the new tissue containment system during laparoscopic ovarian cystectomy. Premenopausal women, aged 18-45 undergoing laparoscopic cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal woman patient age 18-45 years
* Women with regular period
* Women with ovarian neoplasm (size: 3-10cm)
* Laparoscopic surgery required
* Body mass index 18.5-27.9kg/m2
* Subject able to comprehend and give informed consent for participation in this study
* Signed informed consent form

Exclusion Criteria:

* Patient is not considered suitable for a laparoscopic ovarian cystectomy procedure
* The ovaries and pelvic cavity are severely adhered, and the tumor ruptures when free
* Women with Polycystic ovary syndrome
* Baseline AMH less than 0.5ng / mL
* Known to have participated in any other clinical trials or hormone therapy within 3 months
* Women during pregnancy and lactation
* Women in acute stage infection of reproductive system or other parts
* Women combined with severe central nervous system, cardiovascular system, liver and kidney, digestive tract, respiratory system, endocrine metabolism (thyroid disease, Cushing syndrome, hyperprolactinemia) and skeletal muscle system and mental disorders contraindicating laparoscopic surgery
* Women with known or suspected poor compliance who cannot complete the trial
* Those who can not sign the informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
The exposure rate | End of study - approximately two years
  • Exposure is defined as "disruption of the device (using dye leak testing or water testing) or visible tissue dissemination".

SECONDARY OUTCOMES:
The ovarian reserve function | Three months after the surgery
  The ovarian reserve function is reflected by the concentration of anti-mullerian hormone(AMH)
Mean procedure time | Within one week after the surgery
  Mean procedure time will be measured by hour/minutes.
Estimated blood loss during operation | Within one week after the surgery
  Blood loss during operation will be measured by volume (mL)
Rate of Intra- or post-operative complications | Three months after the surgery
  Intra or post complications rate (e.g. urinary, intestinal or nerve injury)
The patients' life quality postoperative: questionaire | Three months after the surgery
  The patients' life quality will be measured by The World Health Organization's Quality of Life Questionnaire-Brief Version（WHOQOL-BREF).The maximum value is 120 and the minimum is 0. The higher score means a better outcome.
The Surgery Task Load Index | Within one week after the surgery
  The Surgery Task Load Index will be measured by questionaire. The maximum value is 120 and the minimum is 0. The higher score means a worse outcome.
The rate of failure during in-bag cystectomy procedure | End of study - approximately two years
  Failure is defined as the operator's inability to successfully insert and extract the device.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China